CLINICAL TRIAL: NCT04372199
Title: VALIDATION OF A SEVERITY SCORE TO IDENTIFY PATIENTS ADMITTED FOR COVID-19 PNEUMONIA AT HIGH RISK FOR AN INTENSIVE APPROACH
Brief Title: SEVERITY SCORE FOR COVID-19 PNEUMONIA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Massimo Montalto, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3112
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-04

CONDITIONS: COVID; Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The outbreak of the coronavirus disease 2019 (COVID-19), first merged in China in December 2019, is now becoming a Public Health Emergency, recently confirmed as a pandemic disease by the World Health Organization.

In particular, since February 2020, a rapidly growing number of cases has been identified in Italy.

The clinical picture of ranges from asymptomatic cases, mild upper respiratory tract infections to severe pneumonia with respiratory failure and death. In most severe cases, COVID-19 disease may be complicated by acute respiratory distress syndrome (ARDS), septic shock and multiorgan failure.

It results fundamental to early identify those subjects who rapidly may worsen their clinical status, often requiring an intensive care unit (ICU) admission.

It has been showed that, mainly in more severe forms of SARS-Cov-2 disease, there is the development of an hyperinflammatory status resembling a cytokine storm syndrome, as already reported in SARS patients.

A recent study by Haung et al. reported that patients with COVID-19 infection showed high amounts of IL1B, IFN-gamma, IP10 and MCP1, probably linked to activated T-helper1 (Th1) cell responses. Those requiring ICU admission had higher levels of cytokines than those subjects not requiring ICU admission, thus suggesting that cytokine storm was associated with disease severity.

A similarity between cytokine profile of COVID-19 disease and secondary haemophagocytic syndrome (sHLH) has been reported. Therefore, it was suggested to screen all patients with severe COVID-19 infection both for hyperinflammatory markers (like ferritin), and the HScore commonly used to generate a probability for diagnosis of sHLH (8), which includes some laboratory parameters like triglycerides, fibrinogen, ferritin, serum aspartate aminostransferase.

Based on our experience on patients affected by pneumonia from Covid19, we have observed that those subjects with a more severe prognosis might have some predictive markers. We intend to verify if these markers can identify those subjects with Covid19 infection who need a more intensive therapy and to find a prognosis score.

ELIGIBILITY:
Inclusion Criteria: Patients with diagnosis of pneumonia, confirmed by chest imaging, Covid-19 test positive

Exclusion Criteria: Age lower than 18 years, pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study sample will be constituted by inpatients cases of COVID-19 admitted to Internal Medicine Department of Fondazione Policlinico A. Gemelli IRCCS.
Sampling Method: Probability Sample
Enrollment: 248 (Estimated)
Dates: Start 2020-04-29 (Actual); Primary Completion 2020-05-27 (Estimated); Study Completion 2020-05-27 (Estimated)

PRIMARY OUTCOMES:
To identify the best predictors of critical coronavirus pneumonia and to realize a simple severity score able to early classify high-risk individuals admitted to Internal Medicine Department for COVID-19 disease, needing an intensive approach | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Massimo Montalto, Roma, Italy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT04372199/Prot_SAP_000.pdf